CLINICAL TRIAL: NCT06466902
Title: Evaluation of Intra-operative Photographs for the Assessment of a Proper Lymphadenectomy in Minimally-invasive Gastric Cancer Surgery (PhotoNodes)
Brief Title: Evaluation of Intra-operative Photographs for the Assessment of a Proper Lymphadenectomy in Minimally-invasive Gastrectomies for Gastric Cancer (PhotoNodes)
Acronym: PhotoNodes
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Federico Marchesi, Associate Professor of General Surgery - University of Parma, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 649/2022/OSS/AOUPR
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Lymphadenectomy; Minimally Invasive Surgery; Gastrectomy for Gastric Cancer; Laparoscopic Surgery; Robotic Surgery; Survival Outcomes; Survival Analysis; Quality Of Care
Keywords: D2 Lymphadenectomy quality assessment; Minimally invasive gastric cancer oncologic surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing minimally invasive gastrectomy: Patients undergoing minimally invasive gastrectomy with D2 lymphadenectomy for gastric cancer
  Interventions: Other: Quality assessment of D2 lymphadenectomy using the PhotoNode Score

INTERVENTIONS:
Other: Quality assessment of D2 lymphadenectomy using the PhotoNode Score — During the surgical procedure, a set of 5 high quality laparoscopic intraoperative images of the surgical field will be put on record. Photographs will be taken at the end of the lymphadenectomy phase, before the reconstructive phase begins.
  Three surgeons will review the images. Quality of D2 lymphadenectomy will be assessed independently rating eight node stations (1, 5, 6, 7, 8a, 9, 11p and 12a), based upon the evaluation of the 5 images. Each node station will be given a score from 0 to 3, corresponding to a judgment of Unevaluable (0), Poor (1), Doubtful (2) or Excellent (3) lymphadenectomy respectively, in that specific node station.
  A total score for each patient will be independently obtained from each reviewer ranging from a minimum of 7 (poor lymphadenectomy) to a maximum of 24 (excellent lymphadenectomy). The PNS for each patient will originate from the average score among the three reviewers.

SUMMARY:
Even after the wide introduction of chemo/radiotherapy in the treatment algorithm, adequate surgery remains the cornerstone of gastric cancer treatment with curative intent. A proper D2 lymphadenectomy is associated with improved cancer specific survival as confirmed in Western countries by fifteen-year follow-up results of Dutch and Italian randomized trials.

In clinical practice, the total number of harvested lymph nodes is often considered as a surrogate marker for adequate D2 lymphadenectomy; nonetheless, the number of retrieved nodes does not necessarily correlate with residual nodes, which intuitively could represent a more reliable marker of surgical adequacy. The availability of an efficient tool for evaluating the absence of residual nodes in the operative field at the end of node dissection could better correlate with survival outcomes.

The goal of this multicentric observational prospective study is to test the reliability of a new score (PhotoNodes Score) created to rate the quality of the lymphadenectomy performed during minimally invasive gastrectomy for gastric cancer. The score is assigned by assessing the absence of residual nodes at the end of node dissection on a set of laparoscopic/robotic high quality intraoperative images collected from each patient undergoing a minimally invasive gastrectomy with D2 node dissection.

Ideally, this tool could be a new indicator of the quality of D2 dissection and could assume a prognostic role in the treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing minimally invasive curative-intent surgery for gastric adenocarcinoma with D2 lymphadenectomy
* Patients undergoing upfront surgery or treated with a neoadjuvant/perioperative chemotherapy
* Total or Subtotal Gastrectomy
* Laparoscopic or Robotic approach

Exclusion Criteria:

* Age less than 18 year old
* Esophago-gastric junction cancer Siewert type I, II or III
* Metastatic disease
* Lymphadenectomy less than D2
* Open surgery
* Conversion to open surgery
* Palliative gastrectomy
* R1 or R2 resection
* Multivisceral resection except for cholecystectomy
* Surgical procedures other than subtotal or total gastrectomy
* A single node station rated as unevaluable by more than one reviewer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing minimally invasive curative-intent surgery for gastric adenocarcinoma with D2 lymphadenectomy at the University Hospital of Parma (Azienda Ospedaliero-Universitaria di Parma, Parma, Italy) and all other hospitals participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
PhotoNode Score interobserver agreement | At the end of enrollment period
  A PhotoNode Score for each patient will be obtained from each reviewer and the interobserver agreement among the reviewers will be analyzed.
  The range of the PhotoNodes Score will go from a minimum of 7 (poor lymphadenectomy) to a maximum of 24 (excellent lymphadenectomy)

SECONDARY OUTCOMES:
Association between PhotoNode Score and disease-free, 1-year and 3-year overall survival | Data for follow up will be extracted through a 6-monthly medical chart review until 3 years after the end of enrollment period
  An average PhotoNode Score for each patient will originate from the average score among the three reviewers. This PhotoNode Score will correlate with clinical endpoints, including disease-free and overall survival.

OTHER OUTCOMES:
Correlation between PhotoNode Score and number of harvested lymph nodes. | 8 weeks after the end of enrollment period
  Any correlation between PNS and number of harvested lymph nodes will also be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Dalmonte, MD, PhD, Study Chair — Azienda Ospedaliero-Universitaria di Parma; Federico Marchesi, Prof., Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (8):
- Italy (8):
  - Ospedale di Cremona - UOC Chirurgia Generale, Cremona, CR
  - Azienda Ospedaliera Universitaria Careggi - Chirurgia dell'Apparato Digerente, Florence, FI
  - Ospedale San Raffaele - Chirurgia Gastroenterologica, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - Policlinico Abano, Abano Terme, PD
  - Azienda Ospedaliera Universitaria Integrata Borgo Trento - Chirurgia Generale ed Esofago Stomaco, Verona, VR
  - Azienda Ospedaliero-Universitaria di Parma, Parma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Jongh C, Triemstra L, van der Veen A, Brosens LA, Nieuwenhuijzen GA, Stoot JH, de Steur WO, Ruurda JP, van Hillegersberg R; LOGICA Study Group. Surgical quality and prospective quality control of the D2-gastrectomy for gastric cancer in the multicenter randomized LOGICA-trial. Eur J Surg Oncol. 2023 Oct;49(10):107018. doi: 10.1016/j.ejso.2023.107018. Epub 2023 Aug 12. PMID 37651889
- [Background] Han SU, Hur H, Lee HJ, Cho GS, Kim MC, Park YK, Kim W, Hyung WJ; Korean Laparoendoscopic Gastrointestinal Surgery Study (KLASS) Group. Surgeon Quality Control and Standardization of D2 Lymphadenectomy for Gastric Cancer: A Prospective Multicenter Observational Study (KLASS-02-QC). Ann Surg. 2021 Feb 1;273(2):315-324. doi: 10.1097/SLA.0000000000003883. PMID 33064386
- [Background] Bencivenga M, Verlato G, Mengardo V, Weindelmayer J, Allum WH. Do all the European surgeons perform the same D2? The need of D2 audit in Europe. Updates Surg. 2018 Jun;70(2):189-195. doi: 10.1007/s13304-018-0542-4. Epub 2018 Jun 4. PMID 29869322
- [Background] de Steur WO, Hartgrink HH, Dikken JL, Putter H, van de Velde CJ. Quality control of lymph node dissection in the Dutch Gastric Cancer Trial. Br J Surg. 2015 Oct;102(11):1388-93. doi: 10.1002/bjs.9891. Epub 2015 Aug 27. PMID 26313463
- [Background] Degiuli M, Reddavid R, Tomatis M, Ponti A, Morino M, Sasako M; of the Italian Gastric Cancer Study Group (IGCSG). D2 dissection improves disease-specific survival in advanced gastric cancer patients: 15-year follow-up results of the Italian Gastric Cancer Study Group D1 versus D2 randomised controlled trial. Eur J Cancer. 2021 Jun;150:10-22. doi: 10.1016/j.ejca.2021.03.031. Epub 2021 Apr 19. PMID 33887514
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Derived] Marchesi F, Valente M, Giacopuzzi S, Baiocchi GL, Morgagni P, Torroni L, Dalmonte G; Italian Research Group for Gastric Cancer (GIRCG). PhotoNodes Protocol: A Multicenter Prospective Study for the Assessment of Proper Lymphadenectomy in Minimally Invasive Gastric Cancer Surgery Using Intraoperative Photographs. Dig Surg. 2025;42(3):146-151. doi: 10.1159/000545846. Epub 2025 Apr 22. PMID 40262552